CLINICAL TRIAL: NCT00814099
Title: Sedation Management in Pediatric Patients With Acute Respiratory Failure
Brief Title: Sedation Management in Pediatric Patients With Acute Respiratory Failure (The RESTORE Study)
Acronym: RESTORE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 611; U01HL086622 (NIH); U01HL086649 (NIH)
Record Dates: First submitted 2008-12-19; First posted 2008-12-23 (Estimated); Last update posted 2015-07-15 (Estimated); Status verified 2015-07

CONDITIONS: Respiratory Insufficiency; Respiratory Distress Syndrome, Newborn; Lung Diseases
Keywords: Acute Respiratory Failure; Acute Lung Injury
MeSH Terms: conditions — Respiratory Insufficiency; Respiratory Distress Syndrome, Newborn; Lung Diseases; Acute Lung Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Participants will receive care at a pediatric ICU that is continuing the usual approach to sedation management.
  Interventions: Behavioral: Usual approach to sedation management
- 2 (Experimental): Participants will receive care at a pediatric ICU that is implementing the team approach to sedation management.
  Interventions: Behavioral: Team approach to sedation management

INTERVENTIONS:
Behavioral: Team approach to sedation management — The team approach to sedation management includes the following:
  * Team education and consensus on the use of sedatives
  * Team identification of the patient's trajectory of illness and daily prescription of a sedation goal
  * A nurse-implemented goal-directed comfort algorithm that guides moment-to-moment titration of opioids and benzodiazepines
  * Team feedback on sedation management performance
  Arms: 2
Behavioral: Usual approach to sedation management — The pediatric ICU will continue its usual approach to sedation management.
  Arms: 1

SUMMARY:
People with acute respiratory failure usually require the use of an artificial breathing machine, known as a mechanical ventilator. Sedative medications, which help keep people calm and reduce anxiety, are often prescribed for children who are on mechanical ventilators. However, the longer that sedative medications are used, the longer a child may need to remain on mechanical ventilation. This study will evaluate the effectiveness of a team approach to sedation management that aims to reduce the number of days that children with acute respiratory failure require mechanical ventilation.

DETAILED DESCRIPTION:
People who are hospitalized for acute respiratory failure are typically supported on mechanical ventilation, which delivers oxygen and a continuous level of pressure to the damaged lungs. Over 90% of infants and children supported on mechanical ventilation receive some form of sedation medication, which helps keep them safe, calm, and comfortable. Unfortunately, the use of sedation medications may prolong the duration of mechanical ventilation, which can lead to an increased risk for pneumonia and other complications.

Recent studies among adults in intensive care units (ICUs) have shown that when doctors and nurses work together as a team to manage the use of sedation medication, patients are taken off mechanical ventilation sooner and with fewer side effects. This team strategy includes the following:

* Training and discussion between doctors and nurses regarding which sedative medications should be used
* Having doctors and nurses jointly identify the patient's progress and a daily sedation medication goal for the patient
* Having nurses use a decision-making tool to help guide changes in a patient's sedative medication dose
* Keeping track of patient care, which allows doctors and nurses to evaluate the effectiveness of how they manage each patient's sedative medication use

This study will examine the use of the sedation management strategy for infants and children in pediatric ICUs who have acute respiratory failure and require mechanical ventilation. The purpose of the study is to evaluate whether this team approach to sedation medication management is more effective than the usual approach at reducing the amount of time children remain on mechanical ventilators. Study researchers will also examine the cost-effectiveness of this approach and associated quality of life factors.

All participants will be enrolled within 24 hours of starting mechanical ventilation and will be monitored until they receive their last dose of sedative medication, hospital discharge, or Day 28 (whichever comes first). During a 3-month baseline period, all participating pediatric ICUs will provide their usual sedation management, and study researchers will review participants' medical records on a daily basis. Each pediatric ICU will then be randomly assigned to either the control group or the team approach group. Pediatric ICUs in the control group will continue to provide usual care for sedation management. Pediatric ICUs in the team approach group will implement the team approach sedation management guidelines. For both groups, pain and sedation levels will be monitored daily, and study researchers will review participants' medical records on a daily basis, too. Six months after hospital discharge, half of the participants and their parents will complete a follow-up survey and take part in a telephone interview to assess quality of life, psychological factors, and health-related resource use.

ELIGIBILITY:
Inclusion Criteria:

* At least 2 weeks of age (and at least 42 weeks post-menstrual age) and less than 18 years of age
* Intubated and mechanically ventilated for acute lung disease

Exclusion Criteria:

* Cyanotic heart disease with unrepaired or palliated right to left intracardiac shunt
* History of single ventricle at any stage of repair
* Congenital diaphragmatic hernia or paralysis
* Primary pulmonary hypertension
* Critical airway or anatomical obstruction of the lower airway
* Ventilator dependent upon pediatric ICU admission
* Neuromuscular respiratory failure
* Spinal cord injury above the lumbar region
* Pain managed by patient-controlled analgesia or epidural catheter
* Patient transferred from an outside ICU where sedatives had already been administered for more than 24 hours
* Family or medical team has decided not to provide full support
* Enrolled in any other critical care interventional clinical trial concurrently or in the 30 days before study entry
* Known allergy to any of the study medications
* Pregnancy

Ages: 2 Weeks to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2449 (Actual)
Dates: Start 2009-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Duration of mechanical ventilation | Measured from the time of endotracheal intubation to the end of scheduled sedation therapy, hospital discharge, or Day 28 (whichever comes first)

SECONDARY OUTCOMES:
Time to recovery of acute respiratory failure | Measured from the time of endotracheal intubation to when participants first meet the criteria to be tested for extubation readiness
Duration of weaning from mechanical ventilation | Measured from the time participants meet the criteria to be tested for extubation readiness until the time of the first successful extubation (defined as extubation for more than 24 hours)
Occurrence of adverse events | Measured for the duration of the study
Detection of life-threatening neurological events | Measured for the duration of the study
Total sedative exposure | Measured for the duration of the study
Occurrence of iatrogenic withdrawal symptoms | Measured for the duration of the study
Pediatric ICU and hospital length of stay | Measured for the duration of the study
Hospital costs | Measured for the duration of the study
Study implementation costs and cost-effectiveness | Measured for the duration of the study
In-hospital mortality | Measured for the duration of the study
Post-discharge quality of life and emotional health | Measured 6 months after pediatric ICU discharge

CONTACTS AND LOCATIONS:
Overall Officials: Martha A.Q. Curley, RN, PhD, Principal Investigator — University of Pennsylvania; David Wypij, PhD, Study Director — Director, Statistics and Data Coordinating Center; Children's Hospital Boston
Locations (31):
- United States (31):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - University Medical Center, The University of Arizona, Tucson, Arizona
  - Children's Hospital and Research Center at Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Salter Packard Children's Hospital at Stanford, Palo Alto, California
  - University of California Davis Medical Center, Sacramento, California
  - Children's Hospital at University of California San Francisco Medical Center, San Francisco, California
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale-New Haven Children's Hospital, New Haven, Connecticut
  - Nemours/Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Holtz Children's Hospital, Miami, Florida
  - Florida Hospital for Children, Orlando, Florida
  - Children's Memorial Hospital, Chicago, Chicago, Illinois
  - Advocate Hope Children's Hospital, Oak Lawn, Illinois
  - University of Maryland Hospital for Children, Baltimore, Maryland
  - Johns Hopkins Children's Center, Baltimore, Maryland
  - University of Massachusetts Memorial Children's Medical Center, Worcester, Massachusetts
  - C. S. Mott Children's Hospital of the University of Michigan, Ann Arbor, Michigan
  - Children's Mercy Hospital, Kansas City, Kansas City, Missouri
  - St. Louis Children's Hospital, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Cohen Children's Medical Center of New York, New Hyde Park, New York
  - The Children's Hospital at Montefiore, The Bronx, New York
  - Duke Children's Hospital and Health Center, Durham, North Carolina
  - Doernbecher Children's Hospital, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Monroe Carell, Jr. Children's Hospital at Vanderbilt, Nashville, Tennessee
  - Medical City Children's Hospital, Dallas, Texas
  - Children's Medical Center Dallas, Dallas, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah

REFERENCES:
- [Derived] Tasker RC. Respiratory Support for Bronchiolitis Management in the PICU: What We Now Know and What We Want to Know. Pediatr Crit Care Med. 2025 Jun 1;26(6):e827-e831. doi: 10.1097/PCC.0000000000003765. Epub 2025 Jun 5. No abstract available. PMID 40471056
- [Derived] Fischer M, Ngendahimana DK, Watson RS, Schwarz AJ, Shein SL. Cognitive, Functional, and Quality of Life Outcomes 6 Months After Mechanical Ventilation for Bronchiolitis: A Secondary Analysis of Data From the Randomized Evaluation of Sedation Titration for Respiratory Failure Trial ( RESTORE ). Pediatr Crit Care Med. 2024 Mar 1;25(3):e129-e139. doi: 10.1097/PCC.0000000000003405. Epub 2023 Dec 1. PMID 38038620
- [Derived] Olszewski AE, Dervan LA, Smith MB, Asaro LA, Wypij D, Curley MAQ, Watson RS. Risk Factors for Positive Post-Traumatic Stress Disorder Screening and Associated Outcomes in Children Surviving Acute Respiratory Failure: A Secondary Analysis of the Randomized Evaluation of Sedation Titration for Respiratory Failure Clinical Trial. Pediatr Crit Care Med. 2023 Mar 1;24(3):222-232. doi: 10.1097/PCC.0000000000003150. Epub 2022 Dec 23. PMID 36728954
- [Derived] Monteiro ACC, Flori H, Dahmer MK, Sim MS, Quasney MW, Curley MAQ, Matthay MA, Sapru A; BALI Study Investigators of the Pediatric Acute Lung Injury and Sepsis Investigators (PALISI) Network. Thrombomodulin is associated with increased mortality and organ failure in mechanically ventilated children with acute respiratory failure: biomarker analysis from a multicenter randomized controlled trial. Crit Care. 2021 Aug 3;25(1):271. doi: 10.1186/s13054-021-03626-1. PMID 34344416
- [Derived] Kopp W, Gedeit RG, Asaro LA, McLaughlin GE, Wypij D, Curley MAQ; Randomized Evaluation of Sedation Titration for Respiratory Failure (RESTORE) Study Investigators. The Impact of Preintubation Noninvasive Ventilation on Outcomes in Pediatric Acute Respiratory Distress Syndrome. Crit Care Med. 2021 May 1;49(5):816-827. doi: 10.1097/CCM.0000000000004819. PMID 33590999
- [Derived] Natale JE, Asaro LA, Joseph JG, Ulysse C, Ascenzi J, Bowens C, Wypij D, Curley MAQ; RESTORE Study Investigators. Association of Race and Ethnicity with Sedation Management in Pediatric Intensive Care. Ann Am Thorac Soc. 2021 Jan;18(1):93-102. doi: 10.1513/AnnalsATS.201912-872OC. PMID 32776853
- [Derived] Curley MAQ, Gedeit RG, Dodson BL, Amling JK, Soetenga DJ, Corriveau CO, Asario LA, Wypij D; RESTORE Investigative Team. Methods in the design and implementation of the Randomized Evaluation of Sedation Titration for Respiratory Failure (RESTORE) clinical trial. Trials. 2018 Dec 17;19(1):687. doi: 10.1186/s13063-018-3075-8. PMID 30558653
- [Derived] Watson RS, Asaro LA, Hertzog JH, Sorce LR, Kachmar AG, Dervan LA, Angus DC, Wypij D, Curley MAQ; RESTORE Study Investigators and the Pediatric Acute Lung Injury and Sepsis Investigators (PALISI) Network. Long-Term Outcomes after Protocolized Sedation versus Usual Care in Ventilated Pediatric Patients. Am J Respir Crit Care Med. 2018 Jun 1;197(11):1457-1467. doi: 10.1164/rccm.201708-1768OC. PMID 29313710
- [Derived] Lebet R, Hayakawa J, Chamblee TB, Tala JA, Singh N, Wypij D, Curley MAQ. Maintaining Interrater Agreement of Core Assessment Instruments in a Multisite Randomized Controlled Clinical Trial: The Randomized Evaluation of Sedation Titration for Respiratory Failure (RESTORE) Trial. Nurs Res. 2017 Jul/Aug;66(4):323-329. doi: 10.1097/NNR.0000000000000224. PMID 28654569
- [Derived] Natale JE, Lebet R, Joseph JG, Ulysse C, Ascenzi J, Wypij D, Curley MAQ; Randomized Evaluation of Sedation Titration for Respiratory Failure (RESTORE) Study Investigators. Racial and Ethnic Disparities in Parental Refusal of Consent in a Large, Multisite Pediatric Critical Care Clinical Trial. J Pediatr. 2017 May;184:204-208.e1. doi: 10.1016/j.jpeds.2017.02.006. Epub 2017 Mar 2. PMID 28410087
- [Derived] Curley MA, Wypij D, Watson RS, Grant MJ, Asaro LA, Cheifetz IM, Dodson BL, Franck LS, Gedeit RG, Angus DC, Matthay MA; RESTORE Study Investigators and the Pediatric Acute Lung Injury and Sepsis Investigators Network. Protocolized sedation vs usual care in pediatric patients mechanically ventilated for acute respiratory failure: a randomized clinical trial. JAMA. 2015 Jan 27;313(4):379-89. doi: 10.1001/jama.2014.18399. PMID 25602358